CLINICAL TRIAL: NCT00578162
Title: A Study of Survivorship Service Capacities Among Health Care Agencies in New York City
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: NYS DEPT HEALTH CANCER SVC PRO (Unknown)
Responsible Party: Sponsor
Other Study IDs: 05-048
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: All Cancers
Keywords: Cancer; Survivors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Data about participating agencies will be collected by electronic survey. Agencies will be identified using the NYSDOH's existing mailing list of care facilities located in the five boroughs of New York City, referral databases and resource guides created by the American Cancer Society (ACS), the New York Hospital Directory.
  Interventions: Behavioral: we will screen potential agencies using our CALL SCRIPT and our AGENCY SCREENER

INTERVENTIONS:
Behavioral: we will screen potential agencies using our CALL SCRIPT and our AGENCY SCREENER — A cancer care facility or 'agency' is the study's unit of analysis. Data about participating agencies will be collected by electronic survey. Agencies will be identified using the NYSDOH's existing mailing list of care facilities located in the five boroughs of New York City, referral databases and resource guides created by the American Cancer Society (ACS), the New York Hospital Directory

SUMMARY:
To describe the range of services available to cancer survivors in the NYC area.

To determine organizations' need for assistance to enhance services for survivors.

DETAILED DESCRIPTION:
To describe the range of services available to cancer survivors in the NYC area.

To determine organizations' need for assistance to enhance services for survivors.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in the study, an agency must:

  1. Be a current provider of either:

     * General health services (GHS), such as primary care, health education and wellness, mental health services, home health care, palliative care, or cancer screening and diagnosis;
     * Cancer-specific medical treatments (CMT), such as cancer surgery, radiation, chemotherapy, hormonal therapy; experimental therapies; cancer pain and symptom management; rehabilitation services; post-treatment monitoring and surveillance; or prophylactic treatments, such as chemoprevention; or
     * Any type of specialized 'post-cancer' or 'after-cancer' medical care or support services (SMC) (i.e., psychotherapeutic, relationship and family, psycho-educational,wellness and quality of life)
  2. Be located within the five boroughs of New York City
  3. Have been serving cancer patients for 12 months or longer, and
  4. Be willing and able to identify an English-speaking representative, 21 years of age or older as its designated key informant.

Exclusion Criteria:

* We will limit this study to provider agencies such as hospitals, diagnostic centers, clinics, health and human service agencies, and grassroots community organizations and public service settings that offer programs for cancer survivors. Independent practitioners or private practice settings will not be surveyed. Our survey questions are intended for major health services organizations and are not appropriate for private practices settings.

We will use our screening questionnaire to determine where or not a given agency should be included or excluded from the study AGENCY SCREENER.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We assume that the collective network of cancer care and support services can be represented with data from no more than 300 New York City agencies, across all five boroughs. Theseagencies would include hospitals, clinical diagnostic centers, and community-based organizations.
Sampling Method: Non-Probability Sample
Dates: Start 2005-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine agencies' need for assistance to enhance services for survivors. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Loundsbury, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Web Site — http://www.mskcc.org